CLINICAL TRIAL: NCT07188831
Title: A Randomized Controlled Trial Examining the Impact of Agarwood Aromatherapy Inhalation on Sleep Quality and Occupational Fatigue in Hospital Staff
Brief Title: Effect of Agarwood (Aquilaria Sinensis) Inhalation Aromatherapy on Workplace Fatigue and Sleep Quality Among Hospital Employees: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Da-Yeh University (Other)
Responsible Party: Principal Investigator, Yi-chen Wu, Assistant Professor, Da-Yeh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DYU-AGARWOOD-2025
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Fatigue; Occupational Stress or Workplace Stress; Sleep Quality
MeSH Terms: conditions — Fatigue; Occupational Stress; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group of agarwood (Experimental): Inhalation of agarwood (Aquilaria crassna, "Guangdong green kyara") wood chips + 2 drops agarwood essential oil in sachet, and exposure during sleep for 7-8 hrs/night × 7 nights
  Interventions: Other: Agarwood Aromatherapy Inhalation
- Group of sachet (Active Comparator): Inhalation of sachet containing diffuser sticks soaked with sweet almond carrier oil (odorless placebo), and same exposure schedule
  Interventions: Other: Agarwood Aromatherapy Inhalation

INTERVENTIONS:
Other: Agarwood Aromatherapy Inhalation — The experimental group will receive agarwood essential oil sachets as the aromatherapy intervention, and participants will place the sachet 60 cm from the nose during sleep for one week.

SUMMARY:
Hospital staff often experience workplace fatigue and poor sleep quality, which can harm their health, reduce job performance, and increase risks to patient safety. Aromatherapy is a simple, non-invasive complementary therapy that may help reduce fatigue and improve sleep. Agarwood (Aquilaria spp.) has calming and relaxing properties, but there is little clinical research on its effectiveness for hospital staff.

This randomized, double-blind, controlled trial will evaluate whether agarwood aromatherapy inhalation can improve fatigue and sleep quality among hospital employees in Taiwan. About 78 participants will be recruited and randomly assigned to one of two groups:

1. Experimental group: Agarwood sachet containing agarwood wood chips and essential oil.
2. Control group: Placebo sachet containing almond oil.

Participants will place the sachet about 60 cm from the nose during sleep for 7 nights. Data will be collected using questionnaires on workplace fatigue and sleep quality (Pittsburgh Sleep Quality Index, PSQI). The main questions this study aims to answer are: 1. Does agarwood aromatherapy reduce workplace fatigue in hospital staff? 2. Does agarwood aromatherapy improve sleep quality compared with placebo?

Findings are expected to provide scientific evidence for using agarwood inhalation as a safe and convenient strategy to improve staff well-being and support a healthier hospital environment.

ELIGIBILITY:
Inclusion Criteria:

* ≥20 years old, hospital employee working ≥30 hrs/week, employed ≥3 months
* Not using sedatives/hypnotics
* Normal olfactory function (verified with coffee/vinegar smell test)
* Clear consciousness, can read and understand Chinese, no major communication barriers
* Not participating in other aromatherapy or relaxation intervention studies

Exclusion Criteria:

* Major psychiatric disorders (e.g., major depression, schizophrenia)
* Malignancy under active radio/chemotherapy
* CNS diseases (e.g., brain tumor)
* History of asthma, fragrance allergy, pregnancy
* Chronic rhinitis, nasal surgery, anosmia
* Permanent night-shift workers (≥ midnight to 5am, as defined by ILO, 1995)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Workplace Fatigue | Baseline and after 1-week intervention
  Change in fatigue levels measured by the Chinese version of the Copenhagen Burnout Inventory (21 items across four domains: personal, work-related, client-related, and overcommitment). Higher scores indicate greater fatigue.

SECONDARY OUTCOMES:
Sleep Quality | Baseline and after 1-week intervention
  Change in sleep quality measured by the Pittsburgh Sleep Quality Index (PSQI, 19 items, 7 domains). Total scores range from 0 to 21, with higher scores indicating poorer sleep quality.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because of privacy concerns and institutional data protection policies.